CLINICAL TRIAL: NCT01406457
Title: Monitoring of Delayed Ischemia After Subarachnoid Hemorrhage
Acronym: MODISH
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Jed Hartings, Research Asst Professor, University of Cincinnati
Other Study IDs: 10-04-21-01
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: No specimens are to be retained.
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal in this research is to develop better ways to detect and treat the damage caused by bleeding in the brain.

DETAILED DESCRIPTION:
Patients who suffer from a bleeding in the brain (stroke or hemorrhage) often experience secondary complications that can occur up to 2 weeks after the initial bleeding. Complications can include decrease of consciousness, weakness or paralysis, difficulty with speech and language, and worsening of brain damage. These decrease a patient's chances for a good recovery. A brain scan will be used to determine the damage caused by the bleeding, and the brain's electrical activity will be monitored to detect abnormal activity. These measures will be analyzed together with routine medical information to better understand and diagnose complications.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years
2. World Federation of Neurosurgery (WFNS) grade III-IV, and grade V patients who improve within 24h after ventriculostomy
3. Diffuse thick or localized thick subarachnoid clot >1 mm on baseline CT (Fisher grade 3-4)
4. Ruptured saccular aneurysm demonstrated by CT-angiography or DSA
5. Onset of aSAH clinical symptoms within the preceding 72h
6. Treatment of aneurysm within 24 h after admission
7. Treatment of aneurysm by clip ligation

Exclusion Criteria:

1. SAH due to other causes (e.g. trauma, fusiform or mycotic aneurysm)
2. Only a thin diffuse layer or no visible subarachnoid blood in the initial CT
3. Admission in a clinical state with unfavourable prognosis (e.g., bilateral dilated, non-reactive pupils for more than 1h)
4. Coagulopathy (thrombocytes <60,000/ml or INR>1.5)
5. Pregnancy
6. Presence of incompatibilities for MRI, such as non-removable metals, artificial joints, electronic devices (pace maker, pumps), etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with subarachnoid hemmorhage clinical symptoms
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed Hartings, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States